CLINICAL TRIAL: NCT02788786
Title: Feasibility and Acceptability of Daily Oral Rinse in Pregnant Women and Impact on Oral Inflammatory Biomarkers in Rural Nepal
Brief Title: Feasibility and Acceptability of Use of Daily Oral Rinse in Pregnant Women in Rural Nepal
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OPP1131701
Record Dates: First submitted 2016-05-24; First posted 2016-06-02 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-01

CONDITIONS: Periodontitis; Premature Birth of Newborn
Keywords: chlorhexidine; cetylpyridinium chloride; gingival crevicular fluid
MeSH Terms: conditions — Periodontitis; Premature Birth | interventions — Chlorhexidine; Cetylpyridinium; Salts; Water

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- chlorhexidine (Experimental): 0.12% w/v chlorhexidine oral rinse; 15ml, twice-daily, for 12 weeks
  Interventions: Drug: Chlorhexidine
- cetylpyridinium chloride (Experimental): non-alcoholic cetylpyridinium chloride oral rinse; 15ml, twice-daily, for 12 weeks
  Interventions: Drug: Cetylpyridinium chloride
- Salt and Water (Active Comparator): Salt and water based oral rinse; 15ml, twice-daily, for 12 weeks
  Interventions: Drug: Salt and Water
- No oral rinse (No Intervention): No rinse provided in this group

INTERVENTIONS:
Drug: Chlorhexidine — non-alcoholic chlorhexidine gluconate antiseptic mouth rinse
  Other Names: chlorhexidine oral rinse
  Arms: chlorhexidine
Drug: Cetylpyridinium chloride — non-alcoholic cetylpyridinium chloride antiseptic mouth rinse
  Arms: cetylpyridinium chloride
Drug: Salt and Water — salt and water mix oral rinse
  Arms: Salt and Water

SUMMARY:
In Nepal, investigators are conducting a cohort study to estimate the relationship between signs of periodontal disease in pregnant women and preterm delivery. Within that cohort study, investigators plan to conduct an individually randomized trial of the acceptability and effect chlorhexidine, cetylpyridinium chloride, and salt water oral rinses on gingival crevicular fluid and plaque during pregnancy. Women for this pilot trial will be chosen from a subset of the area currently engaged in the larger cohort study, to simplify logistics. The pilot trial will have four arms (three oral rinse arms, and one control group).

* Arm 1: Twice daily oral rinse containing chlorhexidine 0.12% w/v (n=25 women with periodontitis
* Arm 2: Twice daily oral rinse with cetylpyridinium chloride (n=50; 25 women with/without periodontitis)
* Arm 3: Twice daily oral rinse with salt and water (n=50: 25 women with/without periodontitis)
* Arm 4: No oral rinse (n=50)

To select and enroll these 175 participants, data collectors will use the information they collected during an oral health clinical examination conducted at the time of enrollment into the broader cohort study; this information will be used to classify women by signs of periodontitis.

Those selected through this above process will be read an additional consent form; those agreeing to participate will be provided with a supply of their assigned rinse (and instructions on its use and handling/storage), or no rinse. Those in the three rinse groups will be asked to use the provided rinse twice per day after brushing and to save the empty bottles for collection by the health care worker. At the end of this first visit, women will additionally provide a venous blood sample to measure systemic inflammation markers and fluoride.

Women receiving the rinse will be visited by study workers periodically to provide more oral rinse and check on their adherence to the rinse. All 175 women will be visited after 12 weeks to undergo a second oral health clinical examination and provide a second set of gingival crevicular fluid and plaque samples, to allow for evaluation of the effect of each of the oral rinses as compared to the normal physiological changes in gingival inflammation and biofilm composition during the course of pregnancy.

At this final visit, the women in the three rinse arms will also answer a short questionnaire to gather feedback on acceptability and adherence to the oral rinse.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant
* <26 weeks gestation at enrollment
* Enrolled in the broader cohort study

Exclusion Criteria:

* Already previously enrolled
* Not Pregnant

Min Age: 15 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2016-06-27 (Actual); Primary Completion 2016-11-15 (Actual); Study Completion 2016-11-15 (Actual)

PRIMARY OUTCOMES:
Acceptability | 12 weeks
  Do women accept the use of their assigned oral rinse?
Inflammatory markers in gingival crevicular fluid (IL-1β, IL-6, IL-10, TNF-α, PGE2, and GM-CSF) | 12 weeks
  Do the oral rinses (or no rinse) have differing impacts on inflammatory markers in gingival crevicular fluid. Specifically, IL-1β, IL-6, IL-10, TNF-α, PGE2, and GM-CSF will be measured (pg/ml) using validated multiplex immunoassays.

CONTACTS AND LOCATIONS:
Overall Officials: Luke C Mullany, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Nepal Nutrition Intervention Project, Hariaun, Sarlahi District, Nepal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Erchick DJ, Rai B, Agrawal NK, Khatry SK, Katz J, LeClerq SC, Reynolds MA, Mullany LC. Oral hygiene, prevalence of gingivitis, and associated risk factors among pregnant women in Sarlahi District, Nepal. BMC Oral Health. 2019 Jan 5;19(1):2. doi: 10.1186/s12903-018-0681-5. PMID 30611255
- [Derived] Lubon AJ, Erchick DJ, Khatry SK, LeClerq SC, Agrawal NK, Reynolds MA, Katz J, Mullany LC. Oral health knowledge, behavior, and care seeking among pregnant and recently-delivered women in rural Nepal: a qualitative study. BMC Oral Health. 2018 Jun 1;18(1):97. doi: 10.1186/s12903-018-0564-9. PMID 29859084